CLINICAL TRIAL: NCT05237804
Title: Evaluation d'Une Intervention Pour Reduire le Delai de Traitement Des Patients Traites Par TAVI
Brief Title: Evaluation of an Intervention to Reduce the Time to Treatment for TAVI Patients
Acronym: TREAT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021/0226/HP
Record Dates: First submitted 2021-12-23; First posted 2022-02-14 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-12

CONDITIONS: Aortic Valve Stenosis
Keywords: Aortic Stenosis; Treatment time; Medico-economy
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: In this study, there is a randomization of the participating centres in 4 groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control group (No Intervention): The randomized centres in this group will not change their practices.
- Patient component (Experimental): The randomized centres in this group will be required to present patients with:
  * A short introductory video, viewed on a tablet during hospitalization for coronary angiography,
  * A paper booklet,
  * A website.
  Interventions: Other: Patient component
- Organisational component (Experimental): The randomized centres in this group will be provided with a list of organisational changes to be implemented to improve patient care times.
  Interventions: Other: Organisational component
- Patient and organisational components (Experimental): The randomized centres in this group will have to implement the two components.
  Interventions: Other: Patient component; Other: Organisational component

INTERVENTIONS:
Other: Patient component — Video, booklet, website
  Arms: Patient and organisational components; Patient component
Other: Organisational component — Coronarography, CT-scan, anesthesia...
  Arms: Organisational component; Patient and organisational components

SUMMARY:
Aortic stenosis (AS) is the most frequent valvulopathy in Western countries. The prevalence of AS is constantly increasing due to the aging of the population. Although significant progress has been made in understanding the pathophysiological mechanisms underlying the onset and progression of AS, there is no medical treatment to slow or prevent its progression. The only treatment available is Aortic Valve Replacement (AVR) performed by surgery or by catheterization (TAVI).

Once a diagnosis has been made and the decision to treat these patients has been taken, the procedure (AVR or TAVI) must be performed rapidly given the poor prognosis of the disease without treatment. Studies have shown that on the waiting list, the probability of death and hospitalisation for heart failure increases with time. This delay could also reduce the effectiveness of TAVI, thus affecting the performance of the healthcare system.

In this study, an intervention combining an e-health component (tool intended for patients, families and health professionals in contact with patients), and an organisational component (for TAVI implanting centres) has been designed. The aim of this study is to evaluate the effectiveness of this intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age;
* Aortic stenosis
* Indication of TAVI
* Patient affiliated or benefiting from a health insurance scheme
* Patient having read and understood the information letter and having signed the consent form

Exclusion Criteria:

* TAVI indication not retained
* Patient who are not fluent in French and have no one around them to translate,
* Patient who do not have access to the Internet (at home or in their immediate environment)
* Proven pregnant woman (positive urine pregnancy test) or breastfeeding or absence of effective contraception (as defined by the WHO) or postmenopausal woman without confirmation diagnosis obtained (amenorrhea not medically induced for at least 12 months before the initiation visit) ;
* Person deprived of their liberty by an administrative or judicial decision or person placed under the protection of justice / guardianship or curators
* History of illness or psychological or sensory abnormality likely to prevent the subject from fully understanding the conditions required for participating in the protocol or preventing him from giving his informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 748 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effectiveness of an intervention combining a patient component and an organisational component | Month 6
  Percentage of patients with a TAVI indication with a time to TAVI procedure of less than 2 months

SECONDARY OUTCOMES:
Time to care, in days | Month 6
  The time to care is the number of days between the date of the initial consultation during which a TAVI is proposed and the date of the TAVI procedure
Mortality rate | Months 3 and 6
  The mortality rate will be measured between the initial consultation during which a TAVI is proposed and the TAVI procedure, and in the three months following the procedure
Patients' health-related quality of life | Baseline, Months 3 and 6
  Patients' health-related quality of life will be measured using the 5-level EQ-5D version (EQ-5D-5L).
Patient knowledge of the disease and the TAVI procedure | Baseline, Month 3
  Patients' knowledge of the disease and the TAVI procedure will be measured by their score to an ad hoc questionnaire (0: minimum score - 26: maximum score).
Medication compliance | Month 6
  Patient medication compliance will be measured using a questionnaire developed by Girerd et al, with a score going from 0 (lowest compliance) to 6 (maximum compliance).
Patient satisfaction | Month 6
  Patient satisfaction with the care they received and (for the group receiving the patient component) with the patient component of the intervention will be measured using a 0 to 10 Likert scale
Number of visits to the patient section of the website | Month 6
  The number of visits to the website will be assessed through Googleanalytics®
Number of visits to the professional section of the website | Month 6
  The number of visits to the website will be assessed through Googleanalytics®
Acceptability of the intervention for participating centers | Month 6
  The acceptability of the intervention will be assessed through an ad hoc questionnaire addressed to TAVI centers and peripheral hospitals performing the coronary angiography of the pre-TAVI assessment.
Intervention components' dose and fidelity | Month 6
  Number of different activities really performed for each component of the intervention / number of activities planned for each component according to the protocol.
Reached populations | Month 6
  Percentage of target individuals who benefit from activities of each component of the intervention
Intervention components' adaptation | Month 6
  Number of activities performed which have been modified to adapt them to the local context / total number of activities performed. A description of the adaptations performed will be provided.
Incremental cost-effectiveness ratio | Month 6
  The incremental cost-effectiveness ratio will be expressed in cost per quality-adjusted life-year (QALY) gained, derived from the EQ-5D-5L questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Helene Eltchaninoff, Pr, Principal Investigator — University Hospital, Rouen
Locations (2):
- France (2):
  - Brest University Hospital, Brest
  - CHU de Rouen, Rouen

IPD SHARING:
Plan to Share IPD: No